CLINICAL TRIAL: NCT02631226
Title: Multi-resistant Enterobacteriaceae Colonisation in Less Than 32 Weeks Pregnant Women Admitted in the Hospital: a Multicenter Study (EME Study).
Brief Title: Multi-resistant Enterobacteriaceae Colonisation in Less Than 32 Weeks Pregnant Women Admitted to the Hospital.
Acronym: EME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Victoria Aldecoa-Bilbao, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: CSPTneonat_2015_01
Record Dates: First submitted 2015-11-30; First posted 2015-12-16 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Multi-resistant Enterobacteriaceae Colonisation; Pregnancy; Nosocomial Outbreaks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pregnant women colonized by resistant enterobacteria

SUMMARY:
The purpose of this study is to determine the prevalence and risk factors for multi-resistant enterobacteriaceae colonization in less than 32 weeks pregnant women admitted to the hospital and its transmission to the newborn, in order to avoid neonatal intensive care unit spread and nosocomial outbreaks.

ELIGIBILITY:
Inclusion Criteria:

* Less than 32 weeks pregnant woman
* Admitted to the hospital

Exclusion Criteria:

* Screening done after 48 hours of admission
* When delivery occurs before screening is performed

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Less than 32 weeks pregnant woman admitted to the hospital and her newborn if the mother is a multi-resistant enterobacteriaceae carrier.
Sampling Method: Non-Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of multi-resistant enterobacteriaceae colonisation in less than 32 weeks pregnant women | 18 months

SECONDARY OUTCOMES:
Prevalence of multi-resistant enterobacteriaceae colonisation of African or Asian pregnant women | 18 months
Incidence of multi-resistant enterobacteriaceae colonisation of pregnant women admitted to the hospital by preterm premature rupture of membranes (PPROM) | 18 months
Transmission rate from the colonized woman to the newborn | 18 months
Number of multi-resisitant enterobacteriacea sepsis in the Neonatal Unit | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Sabadell. Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided